CLINICAL TRIAL: NCT05775497
Title: Optimizing an Online Behavioral Weight Loss Intervention and Novel Culturally Tailored Components for Sexual Minority Women: MOST Optimization Phase
Brief Title: Optimizing an Online Behavioral Weight Loss Intervention and Novel Culturally Tailored Components for Sexual Minority Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1550062-02
Record Dates: First submitted 2023-02-28; First posted 2023-03-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Obesity
Keywords: Sexual minority women; LGBTQ health; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Coping Skills

STUDY DESIGN:
Intervention Model Description: Participants (anticipated n=88) will receive the 12-week online weight loss treatment and will be randomized to receive 0-3 novel intervention components (targeting minority stress, negative body image, and social support). The primary outcome (weight loss) will be assessed at baseline, post-treatment (12 weeks), and follow-up (24 weeks).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Weight Loss Program Only (Experimental): Participants complete an online behavioral weight loss program.
  Interventions: Behavioral: Behavioral weight loss intervention (Online; Rx Weight Loss)
- Weight Loss Program + Coping with Stress Program (Experimental): Participants complete (1) an online behavioral weight loss program and (2) an adjunctive intervention that teaches strategies for coping with stress & stigma due to weight, sexual orientation, and gender & its impact on weight loss.
  Interventions: Behavioral: Behavioral weight loss intervention (Online; Rx Weight Loss); Behavioral: Minority stress intervention
- Weight Loss Program + Coping with Stress Program + Body Image Program (Experimental): Participants complete (1) an online behavioral weight loss program, (2) an adjunctive intervention that teaches strategies for coping with stress & stigma due to weight, sexual orientation, and gender & its impact on weight loss, and (3) an adjunctive intervention for improving negative body image and reducing its impact on weight loss.
  Interventions: Behavioral: Behavioral weight loss intervention (Online; Rx Weight Loss); Behavioral: Minority stress intervention; Behavioral: Negative body image intervention
- Weight Loss Program + Coping with Stress Program + Body Image Program + Social Support Program (Experimental): Participants complete (1) an online behavioral weight loss program, (2) an adjunctive intervention that teaches strategies for coping with stress & stigma due to weight, sexual orientation, and gender & its impact on weight loss, (3) an adjunctive Social Support Intervention that provides participants with online opportunities to give and receive real-time social support for weight loss efforts, and (4) an adjunctive intervention for improving negative body image and reducing its impact on weight loss.
  Interventions: Behavioral: Behavioral weight loss intervention (Online; Rx Weight Loss); Behavioral: Minority stress intervention; Behavioral: Social support intervention; Behavioral: Negative body image intervention
- Weight Loss Program + Body Image Program + Social Support Program (Experimental): Participants complete (1) an online behavioral weight loss program, (2) an adjunctive Social Support Intervention that provides participants with online opportunities to give and receive real-time social support for weight loss efforts, and (3) an adjunctive intervention for improving negative body image and reducing its impact on weight loss.
  Interventions: Behavioral: Behavioral weight loss intervention (Online; Rx Weight Loss); Behavioral: Social support intervention; Behavioral: Negative body image intervention
- Weight Loss Program + Coping with Stress Program + Social Support Program (Experimental): Participants complete a (1) online behavioral weight loss program, (2) an adjunctive intervention that teaches strategies for coping with stress & stigma due to weight, sexual orientation, and gender & its impact on weight loss, and (3) an adjunctive Social Support Intervention that provides participants with online opportunities to give and receive real-time social support for weight loss efforts.
  Interventions: Behavioral: Behavioral weight loss intervention (Online; Rx Weight Loss); Behavioral: Minority stress intervention; Behavioral: Social support intervention
- Weight Loss Program + Body Image Program (Experimental): Participants complete (1) an online behavioral weight loss program and (2) an adjunctive intervention for improving negative body image and reducing its impact on weight loss.
  Interventions: Behavioral: Behavioral weight loss intervention (Online; Rx Weight Loss); Behavioral: Negative body image intervention
- Weight Loss Program + Social Support Program (Experimental): Participants complete (1) an online behavioral weight loss program and (2) an adjunctive Social Support Intervention that provides participants with online opportunities to give and receive real-time social support for weight loss efforts.
  Interventions: Behavioral: Behavioral weight loss intervention (Online; Rx Weight Loss); Behavioral: Social support intervention

INTERVENTIONS:
Behavioral: Behavioral weight loss intervention (Online; Rx Weight Loss) — Rx Weight Loss is a fully automated online behavioral obesity treatment that includes 3 core components: weekly online video lessons, submission of self-monitored weight, calorie intake, and activity data, and personalized automated feedback. Participants set goals for weight loss (e.g., 10%), daily calorie intake, and activity (e.g., 200 mins/week of moderate-to-vigorous intensity physical activity). Online lessons discuss healthy eating, physical activity, and behavioral skills (e.g., stimulus control, goal-setting, problem solving). To maintain participant engagement, lessons are interactive, use audio and video, and include experiential learning opportunities. Based on their progress, participants receive automated feedback that provides encouragement, praise for meeting goals, and constructive feedback. To enhance adherence, participants who do not view the weekly lesson or enter monitoring data receive e-mail reminders to re-engage.
Behavioral: Minority stress intervention — The Minority Stress Intervention will teach cognitive and behavioral strategies for coping with minority stress with a focus on how minority stress impacts weight loss behaviors. The treatment will primarily address stressors due to sexuality and weight but will also cover how minority stress intersects with other facets of identity. The intervention, while innovative, is adapted from evidence-based treatments using cognitive behavioral therapy (CBT) to address minority stress.Lessons will provide psychoeducation on minority stress related to sexuality, gender, and weight, how it intersects with other aspects of identity, and how it can interfere with weight loss (e.g., unhealthy eating, avoiding exercise and healthcare, reduced motivation, disengaging from the program).The treatment will be delivered in 12 8-10-min lessons/week (a duration comparable to previous treatments) viewed directly after Rx Weight Loss lessons in Wks 1-12.
  Other Names: Coping with Stress Program
  Arms: Weight Loss Program + Coping with Stress Program; Weight Loss Program + Coping with Stress Program + Body Image Program; Weight Loss Program + Coping with Stress Program + Body Image Program + Social Support Program; Weight Loss Program + Coping with Stress Program + Social Support Program
Behavioral: Social support intervention — The Social Support Intervention will provide sexual minority women with online opportunities to give and receive real-time social support for weight loss efforts. The treatment is based on Social Learning Theory and evidence-based online social support programs used in behavioral weight loss. The intervention will include one video lesson outlining the value of social support for weight loss and well-being, strategies for eliciting support, and an orientation to using the online platform (hosted within Rx Weight Loss). The platform will feature a private forum where participants can post to provide support and discuss their weight loss goals, challenges, and successes. To foster engagement, discussion topics will be automated to post 4 times/week and those who do not participate will be reminded via e-mail to engage (1x/month).
  Other Names: Social Support Program
  Arms: Weight Loss Program + Body Image Program + Social Support Program; Weight Loss Program + Coping with Stress Program + Body Image Program + Social Support Program; Weight Loss Program + Coping with Stress Program + Social Support Program; Weight Loss Program + Social Support Program
Behavioral: Negative body image intervention — The Negative Body Image Intervention will teach CBT skills for improving negative body image and reducing its impact on weight loss behaviors. The treatment is derived from evidence-based CBT interventions targeting body image for women with obesity during behavioral weight loss and will be adapted to reflect the unique body image ideals and concerns of sexual minority women. Lessons will teach CBT strategies for coping with negative body image and reducing interference with weight loss efforts. The intervention will be delivered in 12 weekly 8-10-minute lessons, a treatment duration comparable to previous treatments and will be viewed immediately following Rx Weight Loss lessons during Weeks 1-12.
  Other Names: Body Image Program
  Arms: Weight Loss Program + Body Image Program; Weight Loss Program + Body Image Program + Social Support Program; Weight Loss Program + Coping with Stress Program + Body Image Program; Weight Loss Program + Coping with Stress Program + Body Image Program + Social Support Program

SUMMARY:
Obesity disproportionately impacts sexual minority women. Behavioral weight loss programs are the gold standard treatment for mild to moderate obesity. The investigators have developed an online behavioral weight loss program that is effective, low-cost, and highly scalable. However, existing research suggests that tailoring treatment to address 3 well-established weight loss barriers in sexual minority women will be critical for maximizing the relevance and efficacy of behavioral weight loss for this group. In the Preparation Phase of this K23, the investigators developed 3 novel treatment components targeting sexual minority women's weight loss barriers (i.e., minority stress, low social support, and negative body image), the investigators piloted the program among sexual minority women of higher weight, and the investigators conducted individual qualitative interviews to elicit feedback on the intervention's acceptability, cultural relevance, usability, and feasibility, and this feedback was used to refine the program.

In the Optimization Phase of this K23 (the current phase), 88 women will receive 12 weeks of Rx Weight Loss and will be randomized to receive 0-3 tailored components in a full factorial design with 23 (8) distinct combinations of components. Novel components that increase mean weight loss (by ≥2%) or the proportion of women achieving clinically meaningful weight loss (by ≥10%) at 6 months will be retained in a finalized obesity treatment package that the investigators will evaluate in a future randomized controlled trial (RCT) (Evaluation Phase). The aims of this study are to:

Aim 2A (Optimization): Use a factorial experiment to determine how 3 novel components impact mean weight loss and the proportion of women achieving a 5+% weight loss at 6 months.

Aim 2B (Mediation): Clarify how tailored components impact weight loss by testing hypothesized mechanisms of action (i.e., coping with stress, perceived social support, weight and shape concerns).

This project will tailor and optimize an evidence-based online behavioral obesity treatment to enhance weight loss outcomes in sexual minority women.

ELIGIBILITY:
* Assigned female at birth and currently identify as female
* Self-identify a minority sexual orientation (e.g.,lesbian, bisexual)
* BMI=25-50kg/m2
* 18-70 years old
* Interested in losing weight
* Regular internet and e-mail access
* No significant weight loss within past 6 months (>5%)
* Fluent in English
* Able to participate in moderate physical activity
* Not currently enrolled in a weight loss program
* Not currently taking weight-loss medication
* Not currently pregnant or trying to get pregnant
* Participated in a previous Phase of this study
* Reports a serious mental/physical health condition that would increase potential risks of treatment to the participant (e.g., active symptoms of psychosis, suicidality, mania, alcohol/substance use, or a medical condition that is serious, active, unstable, and degenerative (e.g., CHF)).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Currently self-identify as female
Enrollment: 88 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Change in Weight | 6 months
  Body weight will be formally assessed by an RA at baseline, 3 months, and 6 months. Mean weight loss from baseline will be calculated.
Proportion of Patients Achieving a Weight Loss of 5+% of Initial Weight | 6 months
  Mean weight loss at 6 months will be used to determine the proportion of participants who achieved clinically significant (5+%) weight loss.

SECONDARY OUTCOMES:
Change in Weight | 3 months
  Body weight will be formally assessed by an RA at baseline, 3 months, and 6 months. Mean weight loss from baseline will be calculated.
Proportion of Patients Achieving a Weight Loss of 5+% of Initial Weight | 3 months
  Mean weight loss at 3 months will be used to determine the proportion of participants who achieved clinically significant (5+%) weight loss.
Change in skills for coping with stress | 3 and 6 months after baseline
  Skills for coping with stress will be measured with the 28-item Brief COPE Scale. This widely used scale assesses adaptive and maladaptive strategies for coping with stress using 14 subscales on a 1 (I havent been doing this at all) to 4 (Ive been doing this a lot) scale. Higher scores represent more frequent coping skill use.
Change in perceived social support | 3 and 6 months after baseline
  Perceived social support will be measured with the 16-item Social Support Behaviors Scale (SSB), which assesses emotional, instrumental, and sexuality-specific social support on a 1-5 scale. Higher scores indicate more support. The SSB shows excellent internal consistency and validity in studies of SGM adults
Change in negative body image | 3 and 6 months after baseline
  Negative body image will be measured with the widely used weight and shape concern subscales of the Eating Disorder Examination Questionnaire. 8 items assess shape concerns and 5 items assess weight concerns on a 0 (not at all) to 6 (markedly) scale.

OTHER OUTCOMES:
Adherence to behavioral weight loss - Online metrics | 3 months after baseline
  There are a number of markers of adherence that tend to be highly correlated and predictive of weight loss success including engagement with the online intervention and number of self-monitoring entries. The investigators will use data collected by the Rx Weight Loss platform to determine the number of lessons viewed, number of self-monitoring data entries, and number of log-ins.
Adherence to behavioral weight loss - Energy intake | 3 months after baseline
  There are a number of markers of adherence that tend to be highly correlated and predictive of weight loss success including daily tracking. Women will self-monitor their daily calorie intake using an app-based program (e.g., MyFitness Pal) and will report their weekly intake weekly in Rx Weight Loss for comparison to their weekly calorie goal.
Adherence to behavioral weight loss - Physical activity | 3 and 6 months after baseline
  Weekly physical activity minutes will be assessed to determine adherence to the goal of 150 minutes of MVPA/week

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Results will be submitted to ClinicalTrials.gov within appropriate timelines. Quantitative data will be published in peer-reviewed manuscripts that will be submitted to PubMed Central upon acceptance.
  Study results will be presented to the scientific community at national conferences relevant to obesity and sexual minority health.
  Aggregate quantitative data may be requested from other researchers 5 years after the completion of the primary endpoint by contacting Dr. Panza. If there are no restrictions imposed by institutional policies, local IRBs, or laws/regulations, the investigators will make de-identified data available to a requester within the context of a clear data-sharing agreement.

DOCUMENTS (1):
  • Informed Consent Form (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT05775497/ICF_000.pdf